CLINICAL TRIAL: NCT06818461
Title: Assessment of Corneal Biomechanical Properties Using Corvis ST Following LASIK, PRK, and CXL
Status: Completed | Type: Observational
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Mohamed Yasser Sayed Saif, Professour of Ophthalmology, Beni-Suef University
Other Study IDs: FMBSUREC/05012025/ Saif
Record Dates: First submitted 2025-02-05; First posted 2025-02-10 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-06

CONDITIONS: Myopia; Keratoconus; Refractive Surgery
Keywords: corneal biomechanics; prk; lasik; cxl
MeSH Terms: conditions — Myopia; Keratoconus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Lasik: a non-contact air puff tonometer combined with Scheimpflug imaging to assess the cornea's deformation response. Measurements will be taken at multiple postoperative time points to track biomechanical changes. Key parameters such as Deformation Amplitude (DA), Stiffness Parameter (SP-A1), Applanation Times (A1 & A2), Peak Distance (PD), and Biomechanically Corrected IOP (bIOP) will be recorded.
  Interventions: Other: Corvis St Before and after lasik, PRK, CXL
- PRK: a non-contact air puff tonometer combined with Scheimpflug imaging to assess the cornea's deformation response. Measurements will be taken at multiple postoperative time points to track biomechanical changes. Key parameters such as Deformation Amplitude (DA), Stiffness Parameter (SP-A1), Applanation Times (A1 & A2), Peak Distance (PD), and Biomechanically Corrected IOP (bIOP) will be recorded.
  Interventions: Other: Corvis St Before and after lasik, PRK, CXL
- CXL: a non-contact air puff tonometer combined with Scheimpflug imaging to assess the cornea's deformation response. Measurements will be taken at multiple postoperative time points to track biomechanical changes. Key parameters such as Deformation Amplitude (DA), Stiffness Parameter (SP-A1), Applanation Times (A1 & A2), Peak Distance (PD), and Biomechanically Corrected IOP (bIOP) will be recorded.
  Interventions: Other: Corvis St Before and after lasik, PRK, CXL

INTERVENTIONS:
Other: Corvis St Before and after lasik, PRK, CXL — corneal biomechanics measurment using corvis St

SUMMARY:
To evaluate corneal biomechanical changes using the Corvis ST in patients who have under-gone LASIK, PRK, and corneal cross-linking (CXL).

DETAILED DESCRIPTION:
This observational study aims to evaluate corneal biomechanical changes in patients who have undergone LASIK, PRK, and corneal cross-linking (CXL) using the Corvis ST (Oculus). A total of 90 patients will be recruited from the ClearVision Laser Center database between January 2025 and December 2025. Participants will undergo non-contact biomechanical assessments at multiple postoperative time points to track corneal stability and elasticity over time.

Data Collection & Measurements Patient demographics, clinical history, and baseline preoperative data, including corneal thickness (pachymetry) and refractive status, will be collected. The Corvis ST will be used to measure key biomechanical parameters, such as Corneal Deformation Amplitude (CDA), Applanation Times (A1T & A2T), Radius of Curvature at Highest Concavity (RHC), Stiffness Parameter (SP-A1), Integrated Radius (IR), and the Corvis Biomechanical Index (CBI).

Measurement Protocol

All measurements will be conducted in a controlled environment with stable room temperature and humidity. Patients will be properly aligned, and three consecutive measurements per eye will be taken to ensure repeatability. Data will be recorded at specific intervals:

LASIK & PRK: 1 month, 3 months, 6 months, and 12 months CXL: 1 month, 3 months, 6 months, 12 months, and 24 months Potential Benefits & Risks The study aims to provide valuable insights into corneal biomechanical stability post-surgery, improving postoperative management and long-term visual outcomes. Risks are minimal, with only transient discomfort associated with the non-invasive Corvis ST measurements.

This study will contribute to a better understanding of corneal biomechanics in refractive and therapeutic procedures, potentially guiding future surgical decisions and patient care strategies.

ELIGIBILITY:
Inclusion Criteria:

- 1. Adults aged 18-60 years. 2. Patients who have undergone LASIK, PRK, or CXL at least 1 month prior to measure-ment.

3. Stable refraction for at least 3 months post-procedure. 4. No evidence of active ocular disease or infection.

Exclusion Criteria:

* 1. History of other ocular surgeries (excluding LASIK, PRK, or CXL). 2. Presence of keratoconus or other corneal ectatic disorders not treated with CXL.

  3. Systemic or ocular conditions affecting corneal biomechanical properties (e.g., dia-betes, connective tissue disorders).

  4. Current or recent use of medications influencing corneal biomechanics.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: patients coming for refractive surgery
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-05-28 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
corneal biomechanics | 6 month

CONTACTS AND LOCATIONS:
Locations (1):
- Clearvision, Mohandessin, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Luce DA. Determining in vivo biomechanical properties of the cornea with an ocular response analyzer. J Cataract Refract Surg. 2005 Jan;31(1):156-62. doi: 10.1016/j.jcrs.2004.10.044. PMID 15721708